CLINICAL TRIAL: NCT00381004
Title: Fludarabine, Cyclophosphamide, and Rituximab (FCR) Plus Sargramostim (GM-CSF) as Frontline Therapy for Symptomatic Chronic Lymphocytic Leukemia
Brief Title: FCR Plus Sargramostim (GM-CSF) as Frontline Therapy for Symptomatic Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0267
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Leukemia; Cyclophosphamide; Fludarabine; Sargramostim; Rituximab; GM-CSF; FCR
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FCR + Sargramostim (Experimental): Fludarabine + Cyclophosphamide + Rituximab (FCR) = Fludarabine - Course 1: 25 mg/m^2 IV Days 2-4; Course 2-6: 25 mg/m^2 IV Days 1-3. Cyclophosphamide - Course 1: 250 mg/m^2 intravenous (IV) Days 2-4; Course 2-6: 250 mg/m^2 Days 1-3. Rituximab - Course 1: 375 mg/m^2 IV over 2-6 hours Day 1; Course 2-6: 500 mg/m^2 IV Day 1. Sargramostim - Course 1: 250 mcg/m^2 subcutaneous (SQ) Days -1 and 5-11; Course 2-6: 250 mcg/m^2 SQ Days -1 and 4-10.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Sargramostim; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — Course 1: 250 mg/m^2 by vein over 5-30 minutes on Days 2, 3, and 4; Course 2 - 6: 250 mg/m^2 by vein over 5-30 minutes on Days 1 - 3
  Other Names: cytoxan; neosar
Drug: Fludarabine — Course 1: 25 mg/m^2 by vein over 5-30 minutes on Days 2,3, and 4; Course 2 - 6: 25 mg/m^2 by vein over 5-30 minutes on Days 1 - 3
  Other Names: Fludarabine monophosphate; Fludara
Drug: Sargramostim — Course 1: 250 mcg/m^2 subcutaneous (SQ) on Days -1 and Days 5 - 11; Course 2 - 6: 250 mcg/m^2 SQ on Days -1 and Days 4 - 10
  Other Names: GM-CSF; Leukine
Drug: Rituximab — Course 1: 375 mg/m^2 by vein over 2-6 Hours on Day 1; Course 2 - 6: 500 mg/m^2 by vein over 2-6 Hours on Day 1
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to learn if using a combination of fludarabine, cyclophosphamide, and rituximab, with sargramostim (GM-CSF) can help to control previously untreated chronic lymphocytic leukemia (CLL). The safety of this combination will also be studied. This study will evaluate antibody-dependent cellular cytotoxicity (ADCC) and its relationship to response.

DETAILED DESCRIPTION:
Fludarabine and cyclophosphamide are designed to enter CLL cells and destroy the "machinery" that allows CLL cells to multiply. Rituximab is designed to bind to CLL cells and cause cell death. GM-CSF is designed to help the bone marrow to produce white cells. It may also increase the target molecule called cluster of differentiation antigen 20 (CD20) for rituximab on the surface of the CLL cells which may improve the activity of rituximab.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete physical exam. Blood (about 2 tablespoons) will be drawn for routine tests. The routine blood draw will include a test for hepatitis B, unless this has been done within the last 6 months. This routine blood draw will also include a pregnancy test for women who are able to have children. To be eligible to take part in this study, the pregnancy test must be negative. A bone marrow aspirate and biopsy will be collected. To collect a bone marrow aspirate and biopsy, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow and bone is withdrawn through a large needle.

If you are found to be eligible to take part in the study, you will receive GM-CSF thorough a needle under your skin on Day 1. Each study cycle is about 4 weeks, but may be longer depending on side effects or leukemia response.

You will receive rituximab through a needle in your vein on Day 2. The first infusion may take up to 8 hours. For every dose of rituximab after that, the infusion may take 2-4 hours. The length of the infusion time depends on whether you have any reactions to the infusion. The dose level of rituximab may be increased for Cycles 2-6 as well. The drugs Tylenol (acetaminophen) and Benadryl (diphenhydramine hydrochloride) will be given before each dose of rituximab. This will be done to decrease the risk of side effects. If side effects do occur during rituximab treatment, the drug may have to be stopped until the side effects go away and then restarted, so your time in the outpatient area may be longer if that occurs.

On Days 3-5 of the first treatment cycle, fludarabine and cyclophosphamide will be given through a needle in your vein. Each infusion will take about 30 minutes. After the first treatment cycle, fludarabine and cyclophosphamide will be given on Days 2, 3, and 4 for every cycle after that.

During each cycle, the day after you receive fludarabine and cyclophosphamide, you will begin to receive GM-CSF. You will receive the drug for 1 week or until your white cell count has returned to an acceptable level.

Cycle 1 will be given at M.D. Anderson's outpatient clinic. In some cases, Cycle 1 may be given in the inpatient area. The other 5 cycles can be given either at M.D. Anderson or at another location.

With the exception of rituximab, the same doses of all other drugs will be used throughout the study unless side effects become severe. In that case, the dose may be lowered, or the treatment may be stopped.

During each cycle, blood (about 1 tablespoon) will be drawn once every 1-2 weeks for routine tests.

You will have a bone marrow biopsy performed at the end of Cycles 3 and 6 to check the status of the disease.

You may remain on study for up to 6 cycles. You will be taken off study if the disease gets worse or if intolerable side effects occur.

Once you are off study, blood (about 2 teaspoons) will be drawn every 6-12 months for routine tests.

This is an investigational study. Fludarabine, cyclophosphamide, rituximab, and GM-CSF are all FDA approved and commercially available. However, their use in this study and in this combination is considered investigational. Up to 60 patients will take part in the study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Untreated CLL, CLL/PLL, or SLL (small lymphocytic lymphoma) with indication for therapy. Indications for therapy include at least one of the following: (1) one or more disease-related symptoms [fever, night sweats, weight loss > 10% in prior 6 months, pronounced fatigue]; (2) advanced stage disease (Rai stage >/= 3 or Binet stage C); (3) autoimmune anemia and/or thrombocytopenia that is unresponsive to other therapies; (4) massive or progressive hepatomegaly and/or splenomegaly and/or lymphadenopathy; (5) recurrent infections; (6) rapid lymphocyte doubling time of < 6 months.
* Patients who have been treated with not more than one regimen of immunotherapy (e.g. rituximab, alemtuzumab, rituximab plus alemtuzumab) for a diagnosis of CLL, CLL/PLL, or SLL (small lymphocytic lymphoma).
* Beta-2-microglobulin </= 4 mg/dL.
* Adequate liver function (total bilirubin </= 2.5 mg/dL, serum glutamate pyruvate transaminase (SGPT) </=4 x ULN) and renal function (serum creatinine </= 2.0 mg/dL and/or creatinine clearance < 30 mL/hour). Patients with renal or liver dysfunction due to suspected organ infiltration by lymphocytes may be eligible after discussion with the Principal Investigator, but upper limits for creatinine even under these circumstances must be creatinine < 3mg/dL and bilirubin < 6 mg/dL. Patients with Gilbert's syndrome may be entered on study with bilirubin levels </= 4 mg/dL.
* Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
* Signed informed consent in keeping with the policies of the hospital.
* Male and female patients who are fertile agree to use an effective barrier method of birth control (ie, latex condom, diaphragm, cervical cap, etc) to avoid pregnancy. Female patients of childbearing potential (non-childbearing is defined as >/= 1 year after menses cease and/or surgically sterilized) need a negative serum or urine pregnancy test within 2 days of study enrollment..

Exclusion Criteria:

* Active hepatitis B (at least one of the following markers positive: HBsAg, hepatitis B e antigen (HBeAg), immunoglobulin M (IgM) anti-HBc, hepatitis B virus (HBV) DNA).
* Concurrent chemotherapy or immunotherapy.
* Pregnant patients.
* History of HIV
* Symptomatic central nervous system (CNS) disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 20, 2006 to June 5, 2008. All recruitment done at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | FCR + Sargramostim
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FCR + Sargramostim
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 55 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Participant Overall Response Rate (ORR) at 6 Months Includes Complete Remissions, Partial Remission, or Nodule Partial Remissions.
Description: Complete Remission:Normal exam/No symptoms; Absolute lymphocyte count (ALC)</=4x10^9/L, Hb>11 g/dL, absolute neutrophil count (ANC)>/=1.5x109/L, & platelet count>100x109/L. Bone marrow:<30% lymphocytes aspirate no biopsy evidence disease; Disappearance palpable lymph nodes/spleen/liver, no new lesions. Partial Remission:ALC reduced 50%,either Hb>11 g/dL or 50% improvement (imp.) in deviation, or ANC>/=1.5x109/L or 50% imp., or platelet>100x109/L or 50% imp. in deviation from normal. Reduced 50% palpable lymph nodes/spleen/liver no new lesions. Nodular Partial Response:ALC</=4x109/L + Hb>11 g/dL, ANC>/=1.5x109/L & platelet count>100x109/L; <30% lymphocytes - bone marrow biopsy aspirate + lymphoid nodules;No palpable lymph nodes/spleen/liver tumors without new lesions. Progressive Disease:50% increase (incr.) ALC>10x109/L twice; tumor lesion incr. 50% over entry or responder size at time max regression &/or appearance new malignant disease; Reappearance bone marrow disease.
Time Frame: Baseline to 6 Months
Measure: Number; unit: Percentage of Participants
Arm/Group | FCR + Sargramostim
Number analyzed (Participants) | 60
Percentage of Participants | 100

2. Secondary Outcome: Number of Participants Progression-free
Description: Participants progression free as measured at six months following start of treatment. Criteria for Progressive Disease (PD): Peripheral blood: 50% increase in ALC with a level > 10 x 109/L on at least 2 occasions 2 weeks apart. Tumor: An increase of a lesion by 50% over the size present at entry on study or for patients who respond, the size at the time of maximum regression and/or the appearance of new areas of malignant disease. Reappearance of bone marrow disease. A deterioration in performance status or increasing symptoms do not constitute disease progression.
Time Frame: 6 months or until disease progression if earlier
Measure: Number; unit: participants
Arm/Group | FCR + Sargramostim
Number analyzed (Participants) | 60
participants | 60

3. Primary Outcome: Number of Participants With Overall Response Includes Complete Remissions, Partial Remission, or Nodule Partial Remissions.
Description: as for outcome 1
Time Frame: Baseline to 6 Months
Measure: Number; unit: Participants
Arm/Group | FCR + Sargramostim
Number analyzed (Participants) | 60
Participants
  Complete Response (CR) | 45
  Nodular Partial Response (nPR) | 6
  Partial Response (PD) | 9

ADVERSE EVENTS:
Time Frame: Adverse event collection through total of 6 courses administered, courses are 28 to 42 days (+/- 7 days) depending on recovery of peripheral blood counts and assessments for toxicities after 3 and 6 courses, up to 252 days.
Arm/Group | FCR + Sargramostim
Serious Adverse Events (participants affected / at risk) | 12/60
Other Adverse Events (participants affected / at risk) | 4/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCR + Sargramostim (N=60)
DEHYDRATION (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DEATH (General disorders) | 1 (1)
FEVER OF UNKNOWN ORIGIN (General disorders) | 1 (1)
FEBRILE NEUTROPENIA (Infections and infestations) | 2 (2)
INFECTION (Infections and infestations) | 2 (2)
SECONDARY MALIGNANCY DUCTAL CARCINOMA IN SITU RIGHT BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SECONDARY MALIGNANCY MDS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
SECONDARY MALIGNANCY SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ENCEPHALOATHY (Nervous system disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCR + Sargramostim (N=60)
Pain/erythema at injection site (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes